CLINICAL TRIAL: NCT01215175
Title: A Multicenter, Double-Blind Study of the Safety, Tolerability, and Immunogenicity of Pneumococcal Conjugate Vaccine (V114) Compared to Prevnar™ in Healthy Adults and Toddlers
Brief Title: Safety and Tolerability Study for the Pneumococcal Conjugate Vaccine V114 Versus Prevnar™ (V114-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-001; 2009-015103-58 (Other: EudraCT Number); V114-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal vaccines
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Prevnar™ - Adult Cohort (Active Comparator): Healthy adult participants received a single 0.5 mL intramuscular injection of Prevnar™ on Day 1.
  Interventions: Biological: Prevnar™
- V114 Adjuvanted -Toddler Cohort (Experimental): Healthy toddler (12-15 months of age) participants who had completed a documented full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of aluminum adjuvanted V114 on Day 1.
  Interventions: Biological: V114, Aluminum Adjuvanted
- V114 Nonadjuvanted-Toddler Cohort (Experimental): Healthy toddlers (12-15 months of age) participants who completed a documented full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of non-adjuvanted V114 on Day 1.
  Interventions: Biological: V114, Aluminum Nonadjuvanted
- Prevnar™- Toddler Cohort (Active Comparator): Healthy toddlers (12-15 months of age) participants who had previously completed a documented full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of Prevnar™ on Day 1.
  Interventions: Biological: Prevnar™
- V114 Adjuvanted -Adult Cohort (Experimental): Healthy adult participants received a single 0.5 mL intramuscular injection of aluminum adjuvanted V114 on Day 1.
  Interventions: Biological: V114, Aluminum Adjuvanted

INTERVENTIONS:
Biological: Prevnar™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg each), serotype 6B (4.4 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose.
  Arms: Prevnar™ - Adult Cohort; Prevnar™- Toddler Cohort
Biological: V114, Aluminum Adjuvanted — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2.0 mcg each), serotype 6B (4.0 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose.
  Arms: V114 Adjuvanted -Adult Cohort; V114 Adjuvanted -Toddler Cohort
Biological: V114, Aluminum Nonadjuvanted — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2.0 mcg each), serotype 6B (4.0 mcg) in each 0.5 mL dose.
  Arms: V114 Nonadjuvanted-Toddler Cohort

SUMMARY:
This study is being conducted to evaluate the safety, tolerability, and immunogenicity of 15-valent pneumococcal conjugate vaccine (V114) compared to Prevnar™ in healthy adults and toddlers.

DETAILED DESCRIPTION:
The study was extended to obtain additional sera from adult participants to support further development, validation, and performance of anti-pneumococcal antibody assays.

ELIGIBILITY:
Inclusion criteria:

Adult Stage:

* Adults ≥18 to 45 years of age in good health.
* Signed and dated informed consent prior to receipt of vaccine.
* Afebrile (<100.4°F [<38.0°C] oral or equivalent) on day of vaccination.
* Participant is able to read, understand, and complete study questionnaires (i.e., the Vaccine Report Card).
* Participant is able to attend all scheduled visits and to comply with the study procedures.
* Participant has access to a telephone.
* Females must have a negative urine pregnancy test.

Toddler Stage:

* Healthy toddlers, 12-15 months of age who have previously completed a documented full 3 dose infant series of Prevnar™ at 2, 4, and 6 months of age.
* Participant's parent/legal guardian understands the study procedures, alternate treatments available and risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
* Afebrile, with a rectal temperature <38.1°C (<100.5°F) or axillary temperature <37.8°C (<100.0°F) on day of vaccination.
* Participant's parent/legal guardian is able to read, understand, and complete study questionnaires (i.e., the Vaccination Report Card).
* Participant is able to attend all scheduled visits and to comply with the study procedures.
* Participant's parent/legal guardian has access to a telephone.

Exclusion criteria:

Adult Stage:

* Receipt of any pneumococcal polysaccharide vaccine at any time or receipt of polysaccharide conjugate vaccine after the second year of life.
* Known hypersensitivity to any component of the pneumococcal conjugate vaccine.
* Known or suspected immunocompromised persons, including persons with congenital immunodeficiency, human immunodeficiency virus (HIV) infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure (most recent serum creatinine values in medical record ≥3 mg/dL), nephritic syndrome, or other conditions associated with immunosuppression such as organ or bone marrow transplant.
* Functional or anatomic asplenia.
* History of autoimmune disease including multiple sclerosis (MS), systemic lupus, polymyositis, inclusion body myositis, dermatomyositis, Hashimoto's thyroiditis, Sjogren's syndrome, rheumatoid arthritis, other autoimmune disorders.
* History of chronic fatigue syndrome.
* Known neurologic or cognitive behavioral disorders including multiple sclerosis (MS), MS-like disease, encephalitis/myelitis, acute disseminating encephalomyelitis (ADEM), pervasive developmental disorder, and related disorders.
* Participant has a coagulation disorder contraindicating IM vaccination.
* Use of any immunosuppressive therapy (Note: topical and inhaled/nebulized steroids are permitted). Participants on corticosteroids should be excluded if they are receiving or are expected to receive, in the period from 30 days prior to Visit 1 through Visit 2, systemic doses greater than required for physiological replacement, i.e., >5 mg of prednisone (or equivalent) daily and for >2 weeks. Excluded immunosuppressive therapies also include chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation, or autoimmune disease.
* Any underlying illness that would complicate evaluation and completion of this study.
* Any licensed non-live virus vaccine administered within the 14 days prior to receipt of study vaccine or is scheduled to receive any other licensed vaccine within 30 days following receipt of study vaccine. (Exception: Inactivated influenza vaccine may be administered during the study, but must be given at least 7 days prior to receipt of the study vaccine or at least 15 days after receipt of the study vaccine.)
* Participant has received a licensed live virus vaccine within 30 days prior of receipt of study vaccine or is scheduled to receive vaccination with a licensed live virus vaccine within 30 days of receipt of study vaccine.
* Participant has received diphtheria toxoid within 6 months prior to receipt of study vaccine.
* Prior receipt of a blood transfusion or blood products including immune globulin administered within the 6 months before receipt of study vaccine.
* Investigational drugs or vaccines received within the 2 months before receipt of study vaccine.
* Participation in another clinical study within 42 days before the beginning or anytime during the duration of the current clinical study.
* Recent hospitalization for acute illness within the 3 months before receipt of study vaccine.
* History of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* History of febrile illness (≥100.40 F [≥38.00 C] oral or equivalent) occurring within 72 hours before receipt of study vaccine.
* Participant is pregnant or breastfeeding or expecting to conceive within the projected duration of the study. Female participants of reproductive potential must have been using 2 acceptable methods of birth control for 2 weeks prior to enrollment, and agree to use 2 acceptable methods of birth control for 1 month after vaccination. (Acceptable methods of birth control include use of hormonal contraceptives, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, tubal ligation, condoms, or abstinence).
* Any participant who cannot be adequately followed for safety according to the protocol plan.
* Participant is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study.
* Any other reason that in the opinion of the investigator may interfere with the evaluation required by the study.

Toddler Stage:

* Have received less than the full 3-dose infant series of Prevnar™ or 3rd dose less than 2 months before study vaccine.
* Known hypersensitivity to any component of the pneumococcal conjugate vaccine.
* Known or suspected impairment of immunological function.
* Participant has a history of congenital or acquired immunodeficiency (e.g., splenomegaly).
* Participant or his/her mother has documented HIV infection.
* Functional or anatomic asplenia.
* History of autoimmune disease including multiple sclerosis (MS), systemic lupus, polymyositis, inclusion body myositis, dermatomyositis, Hashimoto's thyroiditis, Sjogren's syndrome, rheumatoid arthritis, other autoimmune disorders.
* Known neurologic or cognitive behavioral disorders including multiple sclerosis (MS), MS-like disease, encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive developmental disorder, and related disorders.
* Receipt of intramuscular, oral, or intravenous corticosteroid treatment within the 2 weeks prior to vaccination. (Note: Toddlers on topical and inhaled/nebulized steroids may participate in the study.) Use of systemic steroids are only permitted when the participant is receiving less than 2 mg/kg per day of prednisone (or its equivalent), or less than 20 mg/d if they weigh more than 10 kg and are not otherwise immunocompromised.
* Participant has received other licensed non-live vaccines administered within the 14 days before receipt of study vaccine.
* Participant has received a licensed live virus vaccine within 30 days prior of receipt of study vaccine (Exception: Influenza virus vaccine given according to recommended guidelines within 7 days of receiving study vaccine).
* Prior receipt of a blood transfusion or blood products, including immunoglobulins.
* Investigational drugs or vaccines received within the 2 months before receipt of study vaccine.
* Participation in another clinical study within 42 days before the beginning or anytime during the duration of the current clinical study.
* History of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* A recent (<72 hours) febrile illness (rectal temperature ≥38.1°C [≥100.5°F]) occurring within 48 hours before receipt of study vaccine.
* History of failure to thrive.
* Participant has a coagulation disorder contraindicating IM vaccination.
* Participant and his/her mother is documented hepatitis B surface antigen-positive.
* Any toddler who cannot be adequately followed for safety according to the protocol plan.
* Participant's parent/legal guardian is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study.
* Any other reason that in the opinion of the investigator may interfere with the evaluation required by the study.

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2010-04-16 (Actual); Study Completion 2011-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sobanjo-ter Meulen A, Vesikari T, Malacaman EA, Shapiro SA, Dallas MJ, Hoover PA, McFetridge R, Stek JE, Marchese RD, Hartzel J, Watson WJ, Musey LK. Safety, tolerability and immunogenicity of 15-valent pneumococcal conjugate vaccine in toddlers previously vaccinated with 7-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2015 Feb;34(2):186-94. doi: 10.1097/INF.0000000000000516. PMID 25741971
- [Derived] McFetridge R, Meulen AS, Folkerth SD, Hoekstra JA, Dallas M, Hoover PA, Marchese RD, Zacholski DM, Watson WJ, Stek JE, Hartzel JS, Musey LK. Safety, tolerability, and immunogenicity of 15-valent pneumococcal conjugate vaccine in healthy adults. Vaccine. 2015 Jun 4;33(24):2793-9. doi: 10.1016/j.vaccine.2015.04.025. Epub 2015 Apr 23. PMID 25913828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 15 sites in the US and Finland. Of the 60 randomized adult participants only one participant discontinued from the study. Of the 90 randomized toddler participants only one participant discontinued from the study. A total of 150 participants were screened and all were enrolled.
Groups:
- V114 Adjuvanted - Adult Cohort: Healthy adult participants received a single 0.5 mL intramuscular injection of aluminum adjuvanted V114 on Day 1.
- V114 Adjuvanted - Toddler Cohort; V114 Nonadjuvanted-Toddler Cohort: Healthy toddlers (12-15 months of age) participants who completed a full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of aluminum non-adjuvanted V114 on Day 1.
- Prevnar™ - Toddler Cohort: Healthy toddlers (12-15 months of age) participants who had previously completed a full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of Prevnar™ on Day 1.
Period: Overall Study
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Started | 30 | 30 | 33 | 29 | 28
Treated | 30 | 30 | 33 | 29 | 28
Completed | 30 | 29 | 33 | 28 | 28
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized participants receiving study treatment; one toddler participant was enrolled in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort | Total
Number analyzed (Participants) | 30 | 30 | 33 | 29 | 28 | 150
Age, Customized [Count of Participants; unit: Participants]
  < 12 months (enrolled in error) | 0 | 0 | 1 | 0 | 0 | 1
  12 Months | 0 | 0 | 16 | 14 | 11 | 41
  13 Months | 0 | 0 | 3 | 4 | 1 | 8
  14 Months | 0 | 0 | 3 | 4 | 6 | 13
  15 Months | 0 | 0 | 10 | 7 | 10 | 27
  18 to 29 Years | 8 | 8 | 0 | 0 | 0 | 16
  30 to 39 Years | 14 | 15 | 0 | 0 | 0 | 29
  40 to 45 Years | 8 | 7 | 0 | 0 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 21 | 15 | 17 | 82
  Male | 17 | 14 | 12 | 14 | 11 | 68

OUTCOME MEASURES:

1. Primary Outcome: Adult: Percentage of Participants With Any Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Day 14 after vaccination
Population: The analysis population included all randomized participants who received study vaccination and who had available post-treatment safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Percentage of Participants | 93.3 | 83.3
Statistical Analysis 1: Comparison: V114 Adjuvanted - Adult Cohort vs Prevnar™ - Adult Cohort; Test type: Other; Risk Difference (RD) = 10.0, 95% CI [-7.4 to 28.3] — Miettinen & Nurminen method

2. Primary Outcome: Toddler: Percentage of Participants With Any Adverse Event
Description: as for outcome 1
Time Frame: Up to Day 14 after vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Percentage of Participants | 93.9 | 89.3 | 85.7
Statistical Analysis 1: Comparison: V114 Adjuvanted - Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 8.2, 95% CI [-7.9 to 26.6] — Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 Nonadjuvanted-Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 3.6, 95% CI [-15.5 to 22.9] — Miettinen & Nurminen method

3. Primary Outcome: Adult: Percentage of Participants With Any Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to Day 14 after vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 Adjuvanted - Adult Cohort vs Prevnar™ - Adult Cohort; Test type: Other; Risk Difference (RD) = 0.0, 95% CI [-11.5 to 11.5] — Miettinen & Nurminen method

4. Primary Outcome: Toddler: Percentage of Participants With Any Serious Adverse Event
Description: as for outcome 3
Time Frame: Up to Day 14 after vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Percentage of Participants | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 Adjuvanted - Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 0.0, 95% CI [-12.2 to 10.6] — Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 Nonadjuvanted-Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 0.0, 95% CI [-12.3 to 12.3] — Miettinen & Nurminen method

5. Primary Outcome: Adult: Percentage of Participants With Any Vaccine-related Adverse Event
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Relatedness of the AE to study vaccine was determined by the investigator.
Time Frame: Up to Day 14 after vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Percentage of Participants | 93.3 | 83.3
Statistical Analysis 1: Comparison: V114 Adjuvanted - Adult Cohort vs Prevnar™ - Adult Cohort; Test type: Other; Risk Difference (RD) = 10.0, 95% CI [-7.4 to 28.3] — Miettinen & Nurminen method

6. Primary Outcome: Toddler: Percentage of Participants With Any Vaccine-related Adverse Event
Description: as for outcome 5
Time Frame: Up to Day 14 after vaccination
Population: The analysis population included all randomized toddler participants who received study vaccination and who had available post-treatment safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Percentage of Participants | 84.8 | 78.6 | 75.0
Statistical Analysis 1: Comparison: V114 Adjuvanted - Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 9.8, 95% CI [-10.6 to 30.9] — Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 Nonadjuvanted-Toddler Cohort vs Prevnar™ - Toddler Cohort; Test type: Other; Risk Difference (RD) = 3.6, 95% CI [-19.1 to 26.0] — Miettinen & Nurminen method

7. Secondary Outcome: Adult: Percentage of Participants Achieving the Immunoglobulin G (IgG) Serotype-specific Threshold Value of ≥ 0.35μg/mL
Description: Immunoglobulin G (IgG) for the serotypes contained in V114 was determined using an electrochemiluminescence assay.
Time Frame: Day 30 after vaccination
Population: The analysis population included all adult participants who did not have a protocol violation that could have impacted the validity of the antibody responses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Percentage of Participants
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 1 (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 41.7 [22.1 to 63.4]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 3 (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 83.3 [62.6 to 95.3]
  Serotype 4: number analyzed (Participants) | 26 | 23
  Serotype 4 | 100.0 [86.8 to 100.0] | 100.0 [85.2 to 100.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 5 (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 95.8 [78.9 to 99.9]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 6A (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 87.0 [66.4 to 97.2]
  Serotype 6B: number analyzed (Participants) | 26 | 23
  Serotype 6B | 96.2 [80.4 to 99.9] | 87.0 [66.4 to 97.2]
  Serotype 7F(non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 7F(non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 50.0 [29.1 to 70.9]
  Serotype 9V: number analyzed (Participants) | 26 | 23
  Serotype 9V | 100.0 [86.8 to 100.0] | 95.7 [78.1 to 99.9]
  Serotype 14: number analyzed (Participants) | 26 | 23
  Serotype 14 | 100.0 [86.8 to 100.0] | 95.7 [78.1 to 99.9]
  Serotype 18C: number analyzed (Participants) | 26 | 23
  Serotype 18C | 100.0 [86.8 to 100.0] | 95.7 [78.1 to 99.9]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 19A (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 19F: number analyzed (Participants) | 26 | 23
  Serotype 19F | 100.0 [86.8 to 100.0] | 100.0 [85.2 to 100.0]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 22F (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 45.8 [25.6 to 67.2]
  Serotype 23F: number analyzed (Participants) | 26 | 23
  Serotype 23F | 96.2 [80.4 to 99.9] | 100.0 [85.2 to 100.0]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 33F (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 62.5 [40.6 to 81.2]

8. Secondary Outcome: Toddler: Percentage of Participants Achieving the Immunoglobulin G (IgG) Serotype-specific Threshold Value of ≥ 0.35μg/mL
Description: Immunoglobulin G (IgG) for the serotypes contained in V114 was determined using an electrochemiluminescence assay.
Time Frame: Day 30 after vaccination
Population: The analysis population included all toddler participants who did not have a protocol violation that could have impacted the validity of the antibody responses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Percentage of Participants
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 1 (non-Prevnar serotype) | 100.0 [88.4 to 100.0] | 95.7 [78.1 to 99.9] | 0.0 [0.0 to 15.4]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 3 (non-Prevnar serotype) | 93.3 [77.9 to 99.2] | 95.7 [78.1 to 99.9] | 18.2 [5.2 to 40.3]
  Serotype 4: number analyzed (Participants) | 30 | 23 | 22
  Serotype 4 | 93.3 [77.9 to 99.2] | 100.0 [85.2 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 5 (non-Prevnar serotype) | 90.0 [73.5 to 97.9] | 95.7 [78.1 to 99.9] | 68.2 [45.1 to 86.1]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 6A (non-Prevnar serotype) | 96.7 [82.8 to 99.9] | 87.0 [66.4 to 97.2] | 86.4 [65.1 to 97.1]
  Serotype 6B: number analyzed (Participants) | 30 | 23 | 22
  Serotype 6B | 100.0 [88.4 to 100.0] | 95.7 [78.1 to 99.9] | 95.5 [77.2 to 99.9]
  Serotype 7F(non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 7F(non-Prevnar serotype) | 90.0 [73.5 to 97.9] | 100.0 [85.2 to 100.0] | 9.1 [1.1 to 29.2]
  Serotype 9V: number analyzed (Participants) | 30 | 23 | 22
  Serotype 9V | 100.0 [88.4 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 14: number analyzed (Participants) | 30 | 23 | 22
  Serotype 14 | 100.0 [88.4 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 18C: number analyzed (Participants) | 30 | 23 | 22
  Serotype 18C | 86.7 [69.3 to 96.2] | 95.7 [78.1 to 99.9] | 100.0 [84.6 to 100.0]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 19A (non-Prevnar serotype) | 83.3 [65.3 to 94.4] | 95.7 [78.1 to 99.9] | 72.7 [49.8 to 89.3]
  Serotype 19F: number analyzed (Participants) | 30 | 23 | 22
  Serotype 19F | 96.7 [82.8 to 99.9] | 100.0 [85.2 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 22F non-Prevnar serotype): number analyzed (Participants) | 33 | 28 | 26
  Serotype 22F non-Prevnar serotype) | 100.0 [89.4 to 100.0] | 100.0 [87.7 to 100.0] | 3.8 [0.1 to 19.6]
  Serotype 23F: number analyzed (Participants) | 30 | 23 | 22
  Serotype 23F | 100.0 [88.4 to 100.0] | 95.7 [78.1 to 99.9] | 100.0 [84.6 to 100.0]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 33F (non-Prevnar serotype) | 63.3 [43.9 to 80.1] | 69.6 [47.1 to 86.8] | 0.0 [0.0 to 15.4]

9. Secondary Outcome: Adult: Geometric Mean Concentration (GMC) of Pneumococcal Serotype Immunoglobulin G (IgG) Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: Day 30 after vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
µg/mL
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 1 (non-Prevnar serotype) | 7.9 [4.5 to 13.8] | 0.7 [0.5 to 1.0]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 3 (non-Prevnar serotype) | 2.9 [2.0 to 4.3] | 1.1 [0.8 to 1.5]
  Serotype 4: number analyzed (Participants) | 26 | 23
  Serotype 4 | 4.2 [2.6 to 6.9] | 3.4 [2.3 to 5.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 5 (non-Prevnar serotype) | 15.1 [8.3 to 27.5] | 1.8 [1.4 to 2.4]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 6A (non-Prevnar serotype) | 12.4 [6.3 to 24.6] | 4.0 [1.9 to 8.6]
  Serotype 6B: number analyzed (Participants) | 26 | 23
  Serotype 6B | 20.1 [10.9 to 37.2] | 5.9 [2.5 to 13.8]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 7F (non-Prevnar serotype) | 6.8 [3.9 to 12.0] | 0.7 [0.5 to 1.0]
  Serotype 9V: number analyzed (Participants) | 26 | 23
  Serotype 9V | 7.9 [4.8 to 13.2] | 7.4 [4.4 to 12.4]
  Serotype 14: number analyzed (Participants) | 26 | 23
  Serotype 14 | 25.8 [15.8 to 42.0] | 12.5 [6.7 to 23.4]
  Serotype 18C: number analyzed (Participants) | 26 | 23
  Serotype 18C | 14.7 [8.7 to 24.8] | 8.6 [4.5 to 16.7]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 19A (non-Prevnar serotype) | 19.1 [12.7 to 28.8] | 5.8 [3.5 to 9.5]
  Serotype 19F: number analyzed (Participants) | 26 | 23
  Serotype 19F | 12.1 [7.1 to 20.6] | 7.5 [4.5 to 12.7]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 22F (non-Prevnar serotype) | 5.9 [3.8 to 8.9] | 0.7 [0.5 to 1.0]
  Serotype 23F: number analyzed (Participants) | 26 | 23
  Serotype 23F | 11.2 [5.8 to 21.7] | 14.2 [7.8 to 25.9]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 33F (non-Prevnar serotype) | 8.2 [4.8 to 14.1] | 1.1 [0.6 to 2.1]

10. Secondary Outcome: Toddler: Geometric Mean Concentration (GMC) of Pneumococcal Serotype Immunoglobulin G (IgG) Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: Day 30 after vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
µg/mL
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 1 (non-Prevnar serotype) | 3.0 [2.3 to 4.1] | 4.3 [2.8 to 6.6] | 0.1 [0.0 to 0.1]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 3 (non-Prevnar serotype) | 2.2 [1.6 to 3.0] | 2.5 [1.7 to 3.6] | 0.4 [0.3 to 0.5]
  Serotype 4: number analyzed (Participants) | 30 | 23 | 22
  Serotype 4 | 1.5 [1.0 to 2.2] | 2.5 [1.7 to 3.9] | 2.8 [1.9 to 4.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 5 (non-Prevnar serotype) | 1.8 [1.3 to 2.5] | 2.5 [1.8 to 3.5] | 0.7 [0.4 to 1.0]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 6A (non-Prevnar serotype) | 3.5 [2.1 to 6.0] | 2.8 [1.6 to 4.9] | 2.2 [1.1 to 4.6]
  Serotype 6B: number analyzed (Participants) | 30 | 23 | 22
  Serotype 6B | 7.1 [4.8 to 10.6] | 8.2 [5.2 to 12.9] | 7.0 [4.5 to 10.9]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 7F (non-Prevnar serotype) | 2.0 [1.4 to 3.0] | 3.2 [2.2 to 4.6] | 0.1 [0.1 to 0.2]
  Serotype 9V: number analyzed (Participants) | 30 | 23 | 22
  Serotype 9V | 3.3 [2.4 to 4.6] | 4.7 [3.3 to 6.8] | 5.9 [3.6 to 9.9]
  Serotype 14: number analyzed (Participants) | 30 | 23 | 22
  Serotype 14 | 9.4 [6.0 to 14.7] | 10.0 [7.1 to 14.1] | 10.8 [6.1 to 18.8]
  Serotype 18C: number analyzed (Participants) | 30 | 23 | 22
  Serotype 18C | 2.1 [1.4 to 3.1] | 2.7 [1.8 to 4.0] | 3.9 [2.7 to 5.8]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 22
  Serotype 19A (non-Prevnar serotype) | 1.6 [1.1 to 2.4] | 2.3 [1.6 to 3.4] | 1.7 [1.0 to 2.7]
  Serotype 19F: number analyzed (Participants) | 30 | 23 | 22
  Serotype 19F | 1.9 [1.4 to 2.7] | 2.7 [1.9 to 3.7] | 4.2 [2.8 to 6.1]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 33 | 23 | 22
  Serotype 22F (non-Prevnar serotype) | 12.5 [8.7 to 17.8] | 8.8 [6.4 to 12.2] | 0.2 [0.1 to 0.3]
  Serotype 23F: number analyzed (Participants) | 30 | 23 | 22
  Serotype 23F | 4.3 [3.1 to 6.0] | 4.3 [3.0 to 6.2] | 7.1 [4.6 to 10.9]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 33 | 23 | 22
  Serotype 33F (non-Prevnar serotype) | 0.9 [0.6 to 1.5] | 1.1 [0.6 to 1.9] | 0.1 [0.1 to 0.2]

11. Secondary Outcome: Adult: Percentage of Participants Achieving Opsonophagocytic Activity (OPA) ≥1:8
Description: OPA for the serotypes contained in V114 was determined using a Multiplex Opsonophagocytic Assay.
Time Frame: Day 30 after vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Percentage of Participants
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 1 (non-Prevnar serotype) | 92.3 [74.9 to 99.1] | 16.7 [4.7 to 37.4]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 3 (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 69.6 [47.1 to 86.8]
  Serotype 4: number analyzed (Participants) | 26 | 24
  Serotype 4 | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 5 (non-Prevnar serotype) | 92.3 [74.9 to 99.1] | 29.2 [12.6 to 51.1]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 6A (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 91.7 [73.0 to 99.0]
  Serotype 6B: number analyzed (Participants) | 26 | 24
  Serotype 6B | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 6C (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 6C (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 79.2 [57.8 to 92.9]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 26 | 22
  Serotype 7F (non-Prevnar serotype) | 96.2 [80.4 to 99.9] | 68.2 [45.1 to 86.1]
  Serotype 9V: number analyzed (Participants) | 26 | 24
  Serotype 9V | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 14: number analyzed (Participants) | 26 | 24
  Serotype 14 | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 18C: number analyzed (Participants) | 26 | 24
  Serotype 18C | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 19A (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 19F: number analyzed (Participants) | 26 | 24
  Serotype 19F | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 22F (non-Prevnar serotype) | 92.3 [74.9 to 99.1] | 45.8 [25.6 to 67.2]
  Serotype 23F: number analyzed (Participants) | 26 | 24
  Serotype 23F | 100.0 [86.8 to 100.0] | 95.8 [78.9 to 99.9]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 33F (non-Prevnar serotype) | 100.0 [86.8 to 100.0] | 100.0 [85.8 to 100.0]

12. Secondary Outcome: Toddler: Percentage of Participants Achieving Opsonophagocytic Activity (OPA) ≥1:8
Description: OPA for the serotypes contained in V114 was determined using a Multiplex Opsonophagocytic Assay.
Time Frame: Day 30 after vaccination
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Percentage of Participants
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 1 (non-Prevnar serotype) | 96.6 [82.2 to 99.9] | 94.7 [74.0 to 99.9] | 0.0 [0.0 to 15.4]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 21
  Serotype 3 (non-Prevnar serotype) | 100.0 [88.1 to 100.0] | 100 [82.4 to 100] | 81.0 [58.1 to 94.6]
  Serotype 4: number analyzed (Participants) | 29 | 19 | 22
  Serotype 4 | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 5 (non-Prevnar serotype) | 96.6 [82.2 to 99.9] | 100.0 [82.4 to 100.0] | 0.0 [0.0 to 15.4]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 6A (non-Prevnar serotype) | 96.6 [82.2 to 99.9] | 100.0 [82.4 to 100.0] | 95.5 [77.2 to 99.9]
  Serotype 6B: number analyzed (Participants) | 29 | 19 | 21
  Serotype 6B | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [83.9 to 100.0]
  Serotype 6C (non-Prevnar serotype): number analyzed (Participants) | 29 | 18 | 21
  Serotype 6C (non-Prevnar serotype) | 79.3 [60.3 to 92.0] | 77.8 [52.4 to 93.6] | 61.9 [38.4 to 81.9]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 7F (non-Prevnar serotype) | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 50.0 [28.2 to 71.8]
  Serotype 9V: number analyzed (Participants) | 29 | 19 | 22
  Serotype 9V | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 14: number analyzed (Participants) | 29 | 19 | 22
  Serotype 14 | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 18C: number analyzed (Participants) | 29 | 19 | 22
  Serotype 18C | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 19A (non-Prevnar serotype) | 96.6 [82.2 to 99.9] | 89.5 [66.9 to 98.7] | 90.9 [70.8 to 98.9]
  Serotype 19F: number analyzed (Participants) | 29 | 19 | 22
  Serotype 19F | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 22F (non-Prevnar serotype) | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 9.1 [1.1 to 29.2]
  Serotype 23F: number analyzed (Participants) | 29 | 19 | 22
  Serotype 23F | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [84.6 to 100.0]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 33F (non-Prevnar serotype) | 100.0 [88.1 to 100.0] | 100.0 [82.4 to 100.0] | 95.5 [77.2 to 99.9]

13. Secondary Outcome: Adult: Geometric Mean Titer (GMT) of Pneumococcal Serotype-specific Opsonophagocytic Activity (OPA)
Description: OPA for the serotypes contained in V114 was determined using a Multiplex Opsonophagocytic Assay
Time Frame: Day 30 after vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 Adjuvanted - Adult Cohort | Prevnar™ - Adult Cohort
Number analyzed (Participants) | 30 | 30
Titer
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 1 (non-Prevnar serotype) | 471.9 [211.0 to 1055.2] | 3.7 [2.0 to 6.9]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 26 | 23
  Serotype 3 (non-Prevnar serotype) | 357.9 [200.8 to 637.8] | 26.1 [11.3 to 60.4]
  Serotype 4: number analyzed (Participants) | 26 | 24
  Serotype 4 | 9684.2 [7150.8 to 13115.2] | 8928.4 [6237.2 to 12780.7]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 5 (non-Prevnar serotype) | 2405.5 [881.8 to 6562.0] | 8.1 [3.3 to 19.9]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 6A (non-Prevnar serotype) | 21117.8 [13491.5 to 33055.2] | 3475.2 [933.3 to 12939.6]
  Serotype 6B: number analyzed (Participants) | 26 | 24
  Serotype 6B | 21795.1 [12869.3 to 36911.7] | 9073.3 [3475.8 to 23685.6]
  Serotype 6C (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 6C (non-Prevnar serotype) | 10940.7 [5931.6 to 20179.8] | 462.6 [99.1 to 2159.4]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 26 | 22
  Serotype 7F (non-Prevnar serotype) | 11685.4 [4940.8 to 27637.0] | 261.4 [55.4 to 1232.4]
  Serotype 9V: number analyzed (Participants) | 26 | 24
  Serotype 9V | 29321.9 [16598.3 to 51798.8] | 18343.5 [11891.7 to 28295.5]
  Serotype 14: number analyzed (Participants) | 26 | 24
  Serotype 14 | 17469.5 [10512.8 to 29029.7] | 13145.2 [8055.9 to 21449.6]
  Serotype 18C: number analyzed (Participants) | 26 | 24
  Serotype 18C | 12180.6 [7864.0 to 18866.5] | 6287.9 [2731.8 to 14473.4]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 19A (non-Prevnar serotype) | 8458.3 [6267.9 to 11414.2] | 2778.0 [1642.0 to 4700.1]
  Serotype 19F: number analyzed (Participants) | 26 | 24
  Serotype 19F | 4597.9 [3251.1 to 6502.8] | 2665.8 [1243.5 to 5714.9]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 22F (non-Prevnar serotype) | 11404.1 [3689.3 to 35251.2] | 41.2 [9.4 to 180.6]
  Serotype 23F: number analyzed (Participants) | 26 | 24
  Serotype 23F | 8616.0 [4380.2 to 16947.8] | 8664.4 [3134.6 to 23949.3]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 26 | 24
  Serotype 33F (non-Prevnar serotype) | 169577.5 [85502.9 to 336322.5] | 8430.4 [4998.6 to 14218.4]

14. Secondary Outcome: Toddler: Geometric Mean Titer (GMT) of Pneumococcal Serotype-specific Opsonophagocytic Activity (OPA)
Description: OPA for the serotypes contained in V114 was determined using a Multiplex Opsonophagocytic Assay
Time Frame: Day 30 after vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 Adjuvanted - Toddler Cohort | V114 Nonadjuvanted-Toddler Cohort | Prevnar™ - Toddler Cohort
Number analyzed (Participants) | 33 | 28 | 28
Titer
  Serotype 1 (non-Prevnar serotype): number analyzed (Participants) | 30 | 23 | 24
  Serotype 1 (non-Prevnar serotype) | 94.0 [56.1 to 157.4] | 164.3 [68.0 to 397.1] | 2.0 [2.0 to 2.0]
  Serotype 3 (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 21
  Serotype 3 (non-Prevnar serotype) | 438.8 [319.0 to 603.6] | 566.2 [400.5 to 800.5] | 33.8 [16.1 to 71.0]
  Serotype 4: number analyzed (Participants) | 29 | 19 | 22
  Serotype 4 | 2933.4 [1939.9 to 4435.5] | 4360.9 [2893.4 to 6572.6] | 5163.6 [3701.1 to 7203.9]
  Serotype 5 (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 5 (non-Prevnar serotype) | 477.6 [257.8 to 884.8] | 1060.2 [736.4 to 1526.4] | 2.0 [2.0 to 2.0]
  Serotype 6A (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 6A (non-Prevnar serotype) | 2894.0 [1439.5 to 5818.1] | 3880.4 [2365.6 to 6365.1] | 2435.8 [981.1 to 6047.2]
  Serotype 6B: number analyzed (Participants) | 29 | 19 | 21
  Serotype 6B | 6884.6 [4192.9 to 11304.3] | 6673.5 [3871.5 to 11503.5] | 8309.3 [5015.1 to 13767.3]
  Serotype 6C (non-Prevnar serotype): number analyzed (Participants) | 29 | 18 | 21
  Serotype 6C (non-Prevnar serotype) | 534.8 [164.9 to 1734.3] | 459.5 [104.7 to 2016.1] | 171.7 [30.7 to 959.0]
  Serotype 7F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 7F (non-Prevnar serotype) | 12555.7 [8244.6 to 19120.9] | 22607.1 [13359.1 to 38257.1] | 56.0 [12.1 to 258.9]
  Serotype 9V: number analyzed (Participants) | 29 | 19 | 22
  Serotype 9V | 5154.5 [3657.2 to 7264.9] | 5933.3 [4529.8 to 7771.6] | 7435.1 [4567.4 to 12103.1]
  Serotype 14: number analyzed (Participants) | 29 | 19 | 22
  Serotype 14 | 5868.1 [3383.3 to 10177.7] | 4408.6 [3248.8 to 5982.5] | 7954.7 [4394.2 to 14399.9]
  Serotype 18C: number analyzed (Participants) | 29 | 19 | 22
  Serotype 18C | 2119.0 [1378.0 to 3258.5] | 3435.2 [2276.4 to 5183.8] | 3862.0 [2520.1 to 5918.3]
  Serotype 19A (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 19A (non-Prevnar serotype) | 1275.2 [718.3 to 2263.9] | 1223.8 [381.9 to 3922.0] | 378.7 [143.3 to 1000.3]
  Serotype 19F: number analyzed (Participants) | 29 | 19 | 22
  Serotype 19F | 1136.4 [734.7 to 1757.5] | 1117.8 [601.5 to 2077.4] | 2493.4 [1567.5 to 3966.2]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 22F (non-Prevnar serotype) | 6736.5 [4594.7 to 9876.8] | 9382.9 [5336.8 to 16496.5] | 4.1 [1.4 to 12.0]
  Serotype 23F: number analyzed (Participants) | 29 | 19 | 22
  Serotype 23F | 7058.5 [4441.1 to 11218.5] | 6150.7 [3615.1 to 10464.9] | 18352.1 [10464.0 to 32186.3]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 29 | 19 | 22
  Serotype 33F (non-Prevnar serotype) | 48824.6 [30727.9 to 77579.0] | 50461.3 [22905.7 to 111166.1] | 2697.9 [1093.7 to 6655.1]

ADVERSE EVENTS:
Time Frame: Up to 1 month after vaccination
Description: The safety population consisted of all randomized participants who received study vaccination and who had available post-treatment safety data.
Groups:
- PREVNAR™-Adult Cohort: Healthy adult participants received a single 0.5 mL intramuscular injection of Prevnar™ on Day 1.
- V114 Adjuvanted- Toddler Cohort; V114 Nonadjuvanted-toddler Cohort: Healthy toddlers (12-15 months of age) participants who completed a full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of aluminum nonadjuvanted V114 on Day 1.
- PREVNAR™- Toddler Cohort: Healthy toddlers (12-15 months of age) participants who had previously completed a full 3-dose infant series of Prevnar™ received a single 0.5 mL intramuscular injection of Prevnar™ on Day 1.
Arm/Group | V114 Adjuvanted -Adult Cohort | PREVNAR™-Adult Cohort | V114 Adjuvanted- Toddler Cohort | V114 Nonadjuvanted-toddler Cohort | PREVNAR™- Toddler Cohort
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/33 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/33 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 28/30 | 25/30 | 31/33 | 25/28 | 24/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Adjuvanted -Adult Cohort (N=30) | PREVNAR™-Adult Cohort (N=30) | V114 Adjuvanted- Toddler Cohort (N=33) | V114 Nonadjuvanted-toddler Cohort (N=28) | PREVNAR™- Toddler Cohort (N=28)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 14 (14) | 10 (10) | 21 (26) | 18 (20) | 17 (18)
Injection site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 10 (10) | 4 (4) | 15 (15) | 6 (6) | 7 (7)
Injection site haematoma (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site nodule (General disorders) | 8 (8) | 5 (5) | 10 (10) | 3 (3) | 7 (7)
Injection site pain (General disorders) | 27 (27) | 24 (24) | 19 (19) | 16 (16) | 10 (10)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 15 (15) | 7 (7) | 11 (11) | 8 (8) | 6 (6)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 1 (3) | 9 (12) | 2 (3) | 2 (2)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (5) | 1 (1) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 11 (12) | 10 (10) | 8 (8) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Data related to the IgG antibody response of serotype 22F in the toddler samples were considered experimental due to failure of assay validity criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.